CLINICAL TRIAL: NCT04434950
Title: A Longitudinal Study for Promotion and Implementation of Repeated HIV Self-testing With Online Real-time Counseling
Brief Title: Promoting Repeated HIV Self-testing Among MSM in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MSS269R
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Behavior, Health
Keywords: HIV testing; HIV self-testing
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Intervention group
  Interventions: Behavioral: Promoting and implementing repeated HIV self-testing and online real-time counseling

INTERVENTIONS:
Behavioral: Promoting and implementing repeated HIV self-testing and online real-time counseling — At baseline, Month 6 and Month 12, participants will view an online video clip promoting the needs for HIV testing in general and HIV self-testing with online real-time counseling. A free HIV self-testing kit will be sent to participants. An HIVST administrator will provide online real-time pre-test and post-test counseling.

SUMMARY:
In this longitudinal study, we will firstly construct a cohort of HIV negative MSM, who will be exposed to an online video-based intervention promoting HIV testing in general and real-time HIV self-testing with online counselling service (HIVST-online) in particular. Participants will receive intervention at baseline, Month 6 and Month 12.

DETAILED DESCRIPTION:
500 MSM will be recruited via venue-based, online outreach, and NGO referrals. At baseline, Month 6 and Month 12, participants received online intervention promoting HIV testing in general and HIV testing with online real-time counseling service. Free HIV self-testing kits will be mailed to participants at baseline, Month 6 and Month 12. Upon appointment, a testing administrator will provide online real-time pre-test and post-test counseling service for HIV self-testing users.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese speaking men
* ≥18 years old
* Anal intercourse with at least one man in the last six months
* Access to online face-to-face communication tools (e.g., Line, Skype, WhatsApp)

Exclusion Criteria:

* Self-reported to be HIV positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
HIV testing of any type | 14 months
  Taking up any type of HIV testing during the follow-up period

SECONDARY OUTCOMES:
HIV self-testing | 14 months
  Taking up HIV self-testing during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No